CLINICAL TRIAL: NCT06142227
Title: The Effect of Reading a Pictorial Storybook on Children's Fear, Anxiety and Emotional Symptoms Before Dental Treatment: A Randomised Controlled Study
Brief Title: The Effect of Reading a Pictorial Storybook on Children's Fear, Anxiety and Emotional Symptoms Before Dental Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gamze Akay (Other)
Collaborators: Artvin Coruh University (Other)
Responsible Party: Sponsor-Investigator, Gamze Akay, Lecturer, Artvin Coruh University
Organization: Artvin Coruh University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Audio book for children
Record Dates: First submitted 2023-11-16; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dental Fear
Keywords: dental fear; Children; dental anxiety; emotional indicators; pictorial storybook

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine dental treatment will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): Before dental treatment, the child will be read a story book with pictures of the dental clinic.
  Interventions: Other: Reading a Pictorial Storybook

INTERVENTIONS:
Other: Reading a Pictorial Storybook — The pictorial storybook by children will be chosen by child psychologists. The book will be read to children by researcher. The researcher has a fairy tale therapy certificate. The pictorial storybook reading will start 15 minutes before the dental treatment process and will be completed before the treatment process begins.. The pictorial storybook will be read to children only one time.
  Arms: Experimental Group

SUMMARY:
The aim of this study was to determine the effect of reading a picture storybook on children's fear, anxiety and emotional symptoms before dental treatment.

DETAILED DESCRIPTION:
In children with receiving dental treatment will be randomly divided into two groups: picture storybook group and control. Interventions will be applied for only 1 times. While the illustrated storybook is read to the experimental group, no intervention will be applied to the control group. The children will be assessed before, during and after. Fear, anxiety and emotional symptoms due to dental treatment procedure will be evaluated using the Children's Emotional Indicator Scale, Child Anxiety Scale-Stateness and Children's Fear Scale.

ELIGIBILITY:
Inclusion Criteria:

* No audiovisual impairment,
* Being open to communication and
* Must be accompanied by a parent.

Exclusion Criteria:

* Having special needs,
* Having an audio-visual impairment,
* Learning difficulties or mental retardation and
* Children whose parents do not agree to participate in the study.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Demographic Information Form | baseline
  It is a form consisting of a total of 13 questions including the child's age, gender, diagnosis, duration of treatment, number of treatments (How many times did the child come to the clinic?), the status of receiving information about dental treatment and the person who received the information, the education level and occupation of the mother and father, the place where the family lives and the economic situation. It was prepared by the researchers in line with the literature.

SECONDARY OUTCOMES:
Child anxiety Scale-State | baseline
  "Child Anxiety Scale-State" scale developed by Ersig et al. in 2013 measures the state anxiety of children aged 4-10 years. In 2017, Gerceker et al. carried out Turkish validity study for the scale. CAS-S (State) is designed as a thermometer. At the bottom is the bulb chamber, and upward are horizontal lines. Each horizontal line represents a score, and the thermometer has 10 points. The bulb chamber at the bottom is 0 points and indicates that there is no anxiety. It is interpreted as the rise of anxiety as it rises upwards. The peak is worth 10 points and refers to the highest anxiety.

OTHER OUTCOMES:
Child Fear Scale | baseline
  This scale was developed by McMurtry et al. in 2011. In 2018, Gerceker et al. carried out a Turkish validity study for the scale. The scale is aimed at children aged 5-10 years. The facial muscle changes in fearful expressions are drawn by a graphic artist based on photos of frightened faces. In this scale, the child is shown a scale containing five facial expressions that are evaluated between 0 and 4 points. While 0 point refers to no fear; 4 points refers to the highest fear.
The Children's Emotional Indicator Scale | baseline
  The Children's Emotional Indicator Scale (CEAS) was developed by Li and Lopez and its Turkish validity and reliability was conducted by Çimke and Bayat. The scale consists of five categories of observable emotional behaviours (Facial expression, Vocalization, Activity, Interaction, and Level of cooperation). Each category has a value between 1-5. The total score that can be obtained from the scale varies between 5-25. The higher the scores obtained from the scale, the higher the negative emotional indicators. Cronbach's alpha value of the scale was 0.92. In the Turkish validity and reliability study of the scale, Cronbach's alpha value was determined as 0.94.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe TAŞTAN, 3, Study Chair — Artvin Coruh University
Locations (1):
- Artvin Oral and Dental Health Centre, Artvin, Turkey (Türkiye)

REFERENCES:
- [Result] Alsaadoon AM, Sulimany AM, Hamdan HM, Murshid EZ. The Use of a Dental Storybook as a Dental Anxiety Reduction Medium among Pediatric Patients: A Randomized Controlled Clinical Trial. Children (Basel). 2022 Mar 1;9(3):328. doi: 10.3390/children9030328. PMID 35327700
- [Result] Aminabadi NA, Vafaei A, Erfanparast L, Oskouei SG, Jamali Z. Impact of pictorial story on pain perception, situational anxiety and behavior in children: a cognitive-behavioral schema. J Clin Pediatr Dent. 2011 Winter;36(2):127-32. doi: 10.17796/jcpd.36.2.3163251527508338. PMID 22524072